CLINICAL TRIAL: NCT01564342
Title: A Prospective Double-Blind Randomized Clinical Trial Comparing Tap Water Irrigation With Normal Saline for Wound Management
Brief Title: Tap Water Versus Normal Saline for Wound Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1272
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Wound Infection Rate
Keywords: wound irrigation; tap water irrigation; wound infection; wound irrigation solution
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wounds irrigated with sterile normal saline (Other): Patients in this arm had their wounds irrigated with sterile normal saline
  Interventions: Procedure: wound irrigation with study fluid
- wound irrigation with tap water (Other): Patients in the arm had their wounds irrigated with tap water
  Interventions: Procedure: wound irrigation with study fluid

INTERVENTIONS:
Procedure: wound irrigation with study fluid — wounds were either irrigated with sterile normal saline or tap water.

SUMMARY:
This study is designed to compare the infection rates in wounds irrigated with sterile normal saline to those irrigated with chlorinated tap water. The hypothesis is that the wound infection rate subsequent to irrigation with tap water is not significantly different than the infection rate for wounds irrigated with sterile normal saline.

Inclusion criteria are patients older than 1-year of age who present to the emergency department with a soft-tissue laceration requiring repair. Exclusion criteria include patients with any underlying immunocompromising illness, current use of antibiotics, puncture or bite wounds, underlying tendon or bone involvement, or wounds more than nine hours old.

Patients are randomized to have their wounds irrigated either with tap water or sterile normal saline prior to closure, controlling for the volume and irrigation method used. Structured follow-up is completed at 48 hours and 30 days to determine the presence of infection.

The primary outcome measure is the difference in wound infection rates between the two randomized groups.

ELIGIBILITY:
Inclusion Criteria:

• Patients older than 1-year of age, who presented to the ED with an uncomplicated soft-tissue laceration requiring repair.

Exclusion Criteria:

* Diabetes mellitus
* Asplenism
* primary immune disorder
* Mechanical heart valve
* Chronic alcoholism
* Steroid use,
* Antibiotics use
* Immunosuppressive chemotherapy
* Wounds older than 9 hours or from a human or animal bite
* Puncture wounds
* Wounds associated with bone, tendon, or neurovascular injury

Min Age: 12 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 1994-06; Primary Completion 1996-06 (Actual); Study Completion 1996-06 (Actual)

PRIMARY OUTCOMES:
Wound Infection at 48 hours | 48 hours
  The primary outcome for this study is the difference in wound infection rates between the two randomized groups. It is assessed at 48 hours

SECONDARY OUTCOMES:
wound infection manifest at 30 days | 30 days
  patients are again contacted at 30 days after repair of their wound to assess for evidence of delayed or late infections

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States